CLINICAL TRIAL: NCT00075842
Title: The Use Of Valeriana Officinalis (Valerian) In Improving Sleep In Patients Who Are Undergoing Adjuvant Treatment For Cancer" A Phase III Randomized, Placebo-Controlled, Double-Blind Study
Brief Title: (Valerian) for Improving Sleep in Patients With Cancer Receiving Adjuvant Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N01C5; NCI-2011-01604 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000349424 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-01-09; First posted 2004-01-13 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Fatigue; Sleep Disorders; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: sleep disorders; unspecified adult solid tumor, protocol specific; fatigue
MeSH Terms: conditions — Fatigue; Sleep Wake Disorders | interventions — Valeriana extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive oral Valeriana officinalis (Valerian) once daily for 8 weeks.
  Interventions: Dietary Supplement: Valeriana officinalis extract
- Arm II (Placebo Comparator): Patients receive an oral placebo once daily for 8 weeks.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: Valeriana officinalis extract — Given orally
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: The herb Valeriana officinalis (valerian) may promote sleep. It is not yet known whether valerian is effective in improving sleep in patients who are receiving adjuvant therapy for cancer.

PURPOSE: This randomized phase III trial is studying how well valerian improves the quality of sleep in patients who are receiving adjuvant therapy (radiation therapy, chemotherapy, or hormone therapy) for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effect of Valeriana officinalis (Valerian) for improving the quality of sleep in patients with cancer receiving adjuvant therapy.

Secondary

* Determine the safety of this therapy, in terms of frequency and severity of adverse events, in these patients.
* Determine the effect of this therapy on the degree of anxiety, fatigue, and activities of daily living in these patients.

OUTLINE: This is a double-blind, placebo-controlled, randomized, multicenter study. Patients are stratified according to type of adjuvant treatment (radiotherapy vs parenteral chemotherapy vs oral therapy vs combined modality), age (40 and under vs 41 to 55 vs 56 to 70 vs over 70), and numerical analogue scale for sleep difficulty (mildly impaired sleep quality [4-7] vs moderate or severely impaired sleep quality [8-10]). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral Valeriana officinalis (Valerian) once daily for 8 weeks.
* Arm II: Patients receive an oral placebo once daily for 8 weeks. After 8 weeks of treatment, patients in arm I may receive Valeriana officinalis (Valerian) for an additional 8 weeks and patients in arm II may cross over to arm I.

Pittsburgh Sleep Quality Index, functional outcomes of sleep, brief fatigue inventory, and profile of mood states questionnaires are completed at baseline and then at weeks 4, 8, 12, and 16.

After completion of study treatment, patients are followed weekly for 2 weeks.

PROJECTED ACCRUAL: A total of 220 patients (110 per treatment arm) will be accrued for this study within approximately 11-22 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer
* Receiving adjuvant therapy, including any of the following:

  * Radiotherapy
  * Parenteral chemotherapy
  * Oral drugs
  * Hormonal therapy
* Previously resected tumor, microscopic disease, or nodal or margin involvement allowed
* Patients receiving intended curative treatment without future planned surgery (i.e., prostate cancer patients receiving radiotherapy followed by hormonal therapy) are eligible
* Reports difficulty sleeping and seeking therapeutic intervention

  * Defined as a score over 3 on the numerical analogue scale
* No obstructive sleep apnea
* No prior diagnosis of primary insomnia per DSM IV criteria

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* At least 6 months

Hepatic

* SGOT ≤ 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 1.5 times ULN

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No chronic symptom that consistently interrupts sleep (e.g., hot flashes, unmanaged pain, or diarrhea)

PRIOR CONCURRENT THERAPY:

Other

* No prior Valeriana officinalis (Valerian) for sleep
* More than 1 month since other prior prescription sleeping-aid medication
* No concurrent benzodiazepines except as short-term treatment for nausea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2003-08; Primary Completion 2007-03 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Insomnia occurrence by Pittsburg Sleep Inventory at 6 weeks | at 6 weeks

SECONDARY OUTCOMES:
Toxicity by questionnaires weekly and CTC grading every 2 weeks | Up to 2 weeks post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Charles L. Loprinzi, MD, Study Chair — Mayo Clinic
Locations (33):
- United States (33):
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Lichfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota

REFERENCES:
- [Result] Barton DL, Atherton PJ, Bauer BA, Moore DF Jr, Mattar BI, Lavasseur BI, Rowland KM Jr, Zon RT, Lelindqwister NA, Nagargoje GG, Morgenthaler TI, Sloan JA, Loprinzi CL. The use of Valeriana officinalis (Valerian) in improving sleep in patients who are undergoing treatment for cancer: a phase III randomized, placebo-controlled, double-blind study (NCCTG Trial, N01C5). J Support Oncol. 2011 Jan-Feb;9(1):24-31. doi: 10.1016/j.suponc.2010.12.008. PMID 21399726